CLINICAL TRIAL: NCT02730598
Title: Determining Efficacy of the Combined Application of Electrical Stimulated Antagonist Contraction During Walking With Sensory TENS for Increasing Strength and Decreasing Pain in Women With Frequent Knee Symptoms
Brief Title: Combined Application of Electrical Stimulated Antagonist Contraction During Walking (Walking Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Kurume University (Other)
Responsible Party: Principal Investigator, Neil Segal, MD, MS, Professor and Faculty Physiatrist, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003435
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hybrid Training System (HTS) (Experimental): HTS stimulation while walking at a comfortable pace for 30 minutes.
  Interventions: Device: Hybrid Training System (HTS)
- Transcutaneous Electrical Nerve Stimulation (TENS) (Active Comparator): Sensory TENS while walking at a comfortable pace for 30 minutes.
  Interventions: Device: Sensory TENS

INTERVENTIONS:
Device: Hybrid Training System (HTS) — Electrodes (15 cm x 6 cm) will be placed over the quadriceps and electrodes (11 cm x 6 cm) (Sekisui Plastics Co., Tokyo, Japan) will be placed over the hamstrings. Electrical stimulation parameters will be based on a standard Russian waveform in which a 5,000 Hz carrier frequency is modulated at 40 Hz (2.4 ms on, 22.6 ms off) to deliver a rectangular voltage biphasic pulse. Acceleration sensors as a joint motion sensor (EWTS9PD, Home Appliances Development Center Corporate Engineering Division, Appliances Company Panasonic Corporation 2-3-1-2 Noji-higashi,Kusatsu City, Shiga, Japan) is placed on the front of each leg 88mm above the patellar edge. It analyzes the algorithm of each exercise pattern, and stimulates the antagonist of the motion of each bilateral knee joint during exercise. Electrical stimulation intensity will be set to ~50-60% of 1RM based on the subject's tolerance. The subject's tolerance gradually increases, and electrical stimulation intensity is reset every 2 weeks.
  Arms: Hybrid Training System (HTS)
Device: Sensory TENS — The electrical stimulation intensity will be set under the muscle contraction threshold (but at a level at which the subject can perceive as sensory TENS). Electrical stimulation parameters (i.e. waveform and pulse duration) will be the same of HTS, while the amplitude will be lower. The subject will be stimulated using the same device as for HTS.
  Arms: Transcutaneous Electrical Nerve Stimulation (TENS)

SUMMARY:
Osteoarthritis of the knee (KOA) is the most common cause of disability in older adults. Osteoarthritis involves a loss of cartilage, which acts like a cushion between the bones as well as changes in the bones of joints. Once the joint cartilage is gone, the body does not produce new cartilage. Joint damage can contribute to pain. Currently, treatment for pain associated with knee osteoarthritis includes exercise. However, exercise at a medium- to high-intensity level can be problematic for people with knee pain. Because exercise is a common treatment for knee pain but many people experience pain during exercise, researchers hope to find a safer and more effective exercise method to strengthen the muscles around the knee.

Both aerobic exercise and resistance exercise are recommended for the treatment of people with knee pain. However, pain can be a barrier to participating in exercise at a moderate or vigorous intensity. Electrical stimulation of muscles holds potential to allow effective exercise to be completed at tolerable intensities. Transcutaneous electrical nerve stimulation (TENS) is the use of very low electric currents produced by a device to stimulate the nerves, to treat pain. Neuromuscular electrical stimulation (NMES) uses low electrical current to cause muscles to contract.

By doing this study, the investigators hope to learn if a hybrid training system (HTS), using a combination of NMES and walking, is effective in strengthening muscles in people with knee pain, aching or stiffness.

In this pilot study, the investigators will use walking with TENS as conventional exercise.

Randomized controlled trial will be conducted to compare the effect of walking augmented by HTS with walking without HTS. The investigators will evaluate the relative advantages of training that combines HTS with conventional walking exercise on the improvement of muscle strength, physical function, and pain relief in obese women with frequent knee symptoms.

Study Hypotheses: Compared with walking with sensory TENS, walking with HTS will:

* 1 increase quadriceps muscle strength.
* 2 decrease knee pain.

Exploratory Hypotheses:

* 3 improve physical function.
* 4 increase PPT (improve central sensitization).
* 5 improve self-reported quality of life.

DETAILED DESCRIPTION:
Osteoarthritis of the knee (KOA) is the most common cause of disability not only in the United States but also in Japan. KOA is associated with pain, quadriceps weakness, swelling, instability, decline of range of motion, physical function, and quality of life (QOL) (1). In particular, quadriceps weakness may contribute to incident symptomatic and progressive disease (2, 3), cause functional limitations and disability (4) and increase the risk of mortality (5). Both aerobic exercise and resistance exercise are recommended for the treatment of people with knee osteoarthritis (KOA) (6). However, exercise at a moderate or severe intensity is often a problem for people with knee pain or a history of knee injury.

Neuromuscular electrical stimulation (NMES) is widely used as a method to increase muscle strength and improve physical function even at a low-moderate exercise intensity (7). However, NMES effect may prove to be insufficient because the exercise intensity is determined by the electrical stimulation endurance level of the user (7). On the other hand, transcutaneous electrical stimulation, so-called transcutaneous electrical nerve stimulation (TENS), is effective for pain relief (8). Knee pain independently reduced quadriceps strength and activation (9). TENS restores inhibited quadriceps motor function (central and muscle activation) through pain relief (10). Moreover the combined application of electrical stimulation (ES) and volitional contractions (VC) is said to be more effective than ES or VC alone (11). Therefore, a hybrid training system (HTS) that resists the motion of a volitionally contracting agonist muscle using the force generated by its electrically stimulated antagonist (NMES) was developed as a way to combine the application of electrical stimulation and voluntary contraction (12). HTS is a method that eliminates the disadvantages of both volitional exercise and NMES (13). It has been reported that HTS is a new training technique that can increase both muscular strength and muscle mass (12, 13, 14, 15). Recently, HTS is showing promise as a countermeasure for the musculoskeletal disuse of astronauts because the HTS technique can generate exercise resistance within the body even if there is no gravity (1). In addition, HTS can be utilized during many different types of exercise (e.g. knee extension exercise, squat and hip flexion, walking exercise, and cycling exercise) (17, 18). It seems to be more effective for improvement of muscle strength and physical function to combine HTS with easy exercise (e.g. knee extension, walking, and squats) for KOA patients.

The main purpose of exercise therapy for KOA is not only muscular strength improvement (the quadriceps femoris muscle in particular) and but also pain relief (19, 20). Muscular strength improvement protects joints and relieves nociceptive stimulation. However, exercise sometimes increases pain. In addition to the pathological change in articular structures, changes in central pain processing or central sensitization appear to be involved in KOA pain (19). Murphy et al. reported that 36% of a heterogenous sample of patients with hip and KOA demonstrated evidence of central sensitization (22). This finding has been incompletely characterized, but it is necessary to consider central sensitization in the treatment of patients with KOA. From a theoretical perspective, exercise has the potential to treat the process of central sensitization: e.g. exercise activates brain-orchestrated endogenous analgesia (23). An initial bout of high intensity eccentric exercise induces central sensitization, but a repeated round of exercise facilitates inherent protective spinal mechanisms (repeated bout effect) (24). Moreover, ipsilateral resistance exercise may possibly prevent the central sensitization (25). Therefore, a time-contingent approach which implies that the patient does not cease exercise bouts once local pain severity increases is recommended (22). A few reports about the dysfunctional endogenous analgesia for patients with musculoskeletal pain response to aerobic exercise were shown, but neither type of aerobic exercise was able to activate endogenous analgesia (24). At present, there is no report of an exercise method that is effective in central sensitization pain patients. Brain-derived neurotrophic factor (BDNF) belongs to the neurotrophic family of growth factors. The loss of BDNF usually leads to neurodegeneration in these motor centers and eventually results in several severe motor diseases, such as amyotrophic lateral sclerosis, spinocerebellar ataxias, Parkinson's disease, Huntington's disease, as well as vestibular syndrome. These neurotrophic factors (e.g., decreasing brain-derived neurotrophic factor) are promising new avenues for diminishing hyperexcitability of the CNS in central sensitization pain patients (2). Da Graca-Tarrago et al. showed that a 30-minute electrical intramuscular stimulation in osteoarthritis decreased pain, increased the local pain pressure threshold (PPT), and decreased BDNF (27). Gajewska-Wozniak et al. reported that low-threshold electrical stimulation of peripheral nerves to stimulate Ia afferent fibers (proprioceptive signaling) might affect the expression of BDNF in rats (28). HTS is an exercise technique that uses electrically eccentric muscle contraction. Yamaguchi et al. showed that the soleus H-reflex increased after one HTS adversely in conventional resistance exercise (29). This seems to indicate that HTS serves to activate Ia fibers. HTS may affect central sensitization and relieve pain in KOA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 40-70 years
3. Knee symptoms (pain, aching, or stiffness) on most of the last 30 days (categorically defined)
4. Body Mass Index (BMI) 30-45kg/m2

Exclusion Criteria:

1. Resistance training at any time in the last 3 months prior to the study
2. Bilateral knee replacement
3. Lower limb amputation
4. Lower limb surgery in the last 6 months that affects walking ability or ability to exercise
5. Back or hip problems that affect walking ability or ability to exercise
6. Unable to walk without a cane or walker
7. Inflammatory joint or muscle disease such as rheumatoid or psoriatic arthritis or polymyalgia rheumatica
8. Multiple sclerosis or other neurodegenerative disorder
9. Known neuropathy
10. Currently being treated with insulin for diabetes
11. Currently being treated for cancer or having untreated cancer
12. Terminal illness (cannot be cured or adequately treated and there is a reasonable expectation of death in the near future)
13. Peripheral Vascular Disease
14. History of myocardial infarction or stroke in the last year
15. Chest pain during exercise or at rest
16. Use of supplemental oxygen
17. Inability to follow protocol (e.g. lack of ability to attend visits or understand instructions)
18. Staff concern for participant health (such as history of dizziness/faintness or current restrictions on activity)
19. Unable to attend more than 2 days within any 1 week or unable to attend 4 or more sessions during the study
20. Implanted cardiac pacemaker, spinal cord stimulator, baclofen or morphine pump or other implanted electrical device.
21. Dermatitis or skin sensitivity to tape used in the study.
22. Pregnancy

Ages: 39 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muraki S, Akune T, Oka H, En-yo Y, Yoshida M, Saika A, Suzuki T, Yoshida H, Ishibashi H, Tokimura F, Yamamoto S, Nakamura K, Kawaguchi H, Yoshimura N. Association of radiographic and symptomatic knee osteoarthritis with health-related quality of life in a population-based cohort study in Japan: the ROAD study. Osteoarthritis Cartilage. 2010 Sep;18(9):1227-34. doi: 10.1016/j.joca.2010.06.001. Epub 2010 Jul 13. PMID 20633679
- [Background] Segal NA, Glass NA, Felson DT, Hurley M, Yang M, Nevitt M, Lewis CE, Torner JC. Effect of quadriceps strength and proprioception on risk for knee osteoarthritis. Med Sci Sports Exerc. 2010 Nov;42(11):2081-8. doi: 10.1249/MSS.0b013e3181dd902e. PMID 20351594
- [Background] Segal NA, Glass NA, Torner J, Yang M, Felson DT, Sharma L, Nevitt M, Lewis CE. Quadriceps weakness predicts risk for knee joint space narrowing in women in the MOST cohort. Osteoarthritis Cartilage. 2010 Jun;18(6):769-75. doi: 10.1016/j.joca.2010.02.002. Epub 2010 Feb 11. PMID 20188686
- [Background] van Dijk GM, Dekker J, Veenhof C, van den Ende CH; Carpa Study Group. Course of functional status and pain in osteoarthritis of the hip or knee: a systematic review of the literature. Arthritis Rheum. 2006 Oct 15;55(5):779-85. doi: 10.1002/art.22244. PMID 17013827
- [Background] Nuesch E, Dieppe P, Reichenbach S, Williams S, Iff S, Juni P. All cause and disease specific mortality in patients with knee or hip osteoarthritis: population based cohort study. BMJ. 2011 Mar 8;342:d1165. doi: 10.1136/bmj.d1165. PMID 21385807
- [Background] Linda S Pescatello, Ross Arena, Deborah Riebe, Paul D Thompson. ACSM's Guidelines for Exercise Testing and Prescription by American College of Sports Medicine., 9nd ed., Wolters Kluwer/Lippincott Williams & Wilkins, Philadelphia, PA. 2014
- [Background] Giggins O, Fullen B, Coughlan G. Neuromuscular electrical stimulation in the treatment of knee osteoarthritis: a systematic review and meta-analysis. Clin Rehabil. 2012 Oct;26(10):867-81. doi: 10.1177/0269215511431902. Epub 2012 Feb 9. PMID 22324059
- [Background] Rutjes AW, Nuesch E, Sterchi R, Kalichman L, Hendriks E, Osiri M, Brosseau L, Reichenbach S, Juni P. Transcutaneous electrostimulation for osteoarthritis of the knee. Cochrane Database Syst Rev. 2009 Oct 7;2009(4):CD002823. doi: 10.1002/14651858.CD002823.pub2. PMID 19821296
- [Background] Park J, Hopkins JT. Induced anterior knee pain immediately reduces involuntary and voluntary quadriceps activation. Clin J Sport Med. 2013 Jan;23(1):19-24. doi: 10.1097/JSM.0b013e3182717b7b. PMID 23103783
- [Background] Son SJ, Kim H, Seeley MK, Feland JB, Hopkins JT. Effects of transcutaneous electrical nerve stimulation on quadriceps function in individuals with experimental knee pain. Scand J Med Sci Sports. 2016 Sep;26(9):1080-90. doi: 10.1111/sms.12539. Epub 2015 Sep 8. PMID 26346597
- [Background] Paillard T. Combined application of neuromuscular electrical stimulation and voluntary muscular contractions. Sports Med. 2008;38(2):161-77. doi: 10.2165/00007256-200838020-00005. PMID 18201117
- [Background] Yanagi T, Shiba N, Maeda T, Iwasa K, Umezu Y, Tagawa Y, Matsuo S, Nagata K, Yamamoto T, Basford JR. Agonist contractions against electrically stimulated antagonists. Arch Phys Med Rehabil. 2003 Jun;84(6):843-8. doi: 10.1016/s0003-9993(02)04948-1. PMID 12808536
- [Background] Matsuse H, Shiba N, Umezu Y, Nago T, Tagawa Y, Kakuma T, Nagata K, Basford JR. Muscle training by means of combined electrical stimulation and volitional contraction. Aviat Space Environ Med. 2006 Jun;77(6):581-5. PMID 16780234
- [Background] Iwasaki T, Shiba N, Matsuse H, Nago T, Umezu Y, Tagawa Y, Nagata K, Basford JR. Improvement in knee extension strength through training by means of combined electrical stimulation and voluntary muscle contraction. Tohoku J Exp Med. 2006 May;209(1):33-40. doi: 10.1620/tjem.209.33. PMID 16636520
- [Background] Takano Y, Haneda Y, Maeda T, Sakai Y, Matsuse H, Kawaguchi T, Tagawa Y, Shiba N. Increasing muscle strength and mass of thigh in elderly people with the hybrid-training method of electrical stimulation and volitional contraction. Tohoku J Exp Med. 2010 May;221(1):77-85. doi: 10.1620/tjem.221.77. PMID 20453461
- [Background] Shiba N, Matsuse H, Takano Y, Yoshimitsu K, Omoto M, Hashida R, Tagawa Y, Inada T, Yamada S, Ohshima H. Electrically Stimulated Antagonist Muscle Contraction Increased Muscle Mass and Bone Mineral Density of One Astronaut - Initial Verification on the International Space Station. PLoS One. 2015 Aug 21;10(8):e0134736. doi: 10.1371/journal.pone.0134736. eCollection 2015. PMID 26296204
- [Background] Matsuse H, Shiba N, Takano Y, Yamada S, Ohshima H, Tagawa Y. Cycling exercise to resist electrically stimulated antagonist increases oxygen uptake in males: pilot study. J Rehabil Res Dev. 2013;50(4):545-54. doi: 10.1682/jrrd.2012.04.0067. PMID 23934874
- [Background] Omoto M, Matsuse H, Takano Y, Yamada S, Ohshima H, Tagawa Y, Shiba N. Oxygen Uptake during Aerobic Cycling Exercise Simultaneously Combined with Neuromuscular Electrical Stimulation of Antagonists. J Nov Physiother. 3-6, 2013.
- [Background] Aguiar GC, Do Nascimento MR, De Miranda AS, Rocha NP, Teixeira AL, Scalzo PL. Effects of an exercise therapy protocol on inflammatory markers, perception of pain, and physical performance in individuals with knee osteoarthritis. Rheumatol Int. 2015 Mar;35(3):525-31. doi: 10.1007/s00296-014-3148-2. Epub 2014 Oct 10. PMID 25300730
- [Background] Vincent KR, Vincent HK. Resistance exercise for knee osteoarthritis. PM R. 2012 May;4(5 Suppl):S45-52. doi: 10.1016/j.pmrj.2012.01.019. PMID 22632702
- [Background] Lluch Girbes E, Nijs J, Torres-Cueco R, Lopez Cubas C. Pain treatment for patients with osteoarthritis and central sensitization. Phys Ther. 2013 Jun;93(6):842-51. doi: 10.2522/ptj.20120253. Epub 2013 Feb 7. PMID 23392185
- [Background] Murphy SL, Lyden AK, Phillips K, Clauw DJ, Williams DA. Subgroups of older adults with osteoarthritis based upon differing comorbid symptom presentations and potential underlying pain mechanisms. Arthritis Res Ther. 2011 Aug 24;13(4):R135. doi: 10.1186/ar3449. PMID 21864381
- [Background] Nijs J, Kosek E, Van Oosterwijck J, Meeus M. Dysfunctional endogenous analgesia during exercise in patients with chronic pain: to exercise or not to exercise? Pain Physician. 2012 Jul;15(3 Suppl):ES205-13. PMID 22786458
- [Background] Hosseinzadeh M, Andersen OK, Arendt-Nielsen L, Madeleine P. Pain sensitivity is normalized after a repeated bout of eccentric exercise. Eur J Appl Physiol. 2013 Oct;113(10):2595-602. doi: 10.1007/s00421-013-2701-0. Epub 2013 Aug 7. PMID 23922170
- [Background] Hosseinzadeh M, Samani A, Andersen OK, Nosaka K, Arendt-Nielsen L, Madeleine P. Ipsilateral resistance exercise prevents exercise-induced central sensitization in the contralateral limb: a randomized controlled trial. Eur J Appl Physiol. 2015 Nov;115(11):2253-62. doi: 10.1007/s00421-015-3205-x. Epub 2015 Jun 24. PMID 26105529
- [Background] Nijs J, Malfliet A, Ickmans K, Baert I, Meeus M. Treatment of central sensitization in patients with 'unexplained' chronic pain: an update. Expert Opin Pharmacother. 2014 Aug;15(12):1671-83. doi: 10.1517/14656566.2014.925446. Epub 2014 Jun 15. PMID 24930805
- [Background] da Graca-Tarrago M, Deitos A, Patricia Brietzke A, Torres IL, Cadore Stefani L, Fregni F, Caumo W. Electrical Intramuscular Stimulation in Osteoarthritis Enhances the Inhibitory Systems in Pain Processing at Cortical and Cortical Spinal System. Pain Med. 2016 May 1;17(5):877-891. doi: 10.1111/pme.12930. Epub 2015 Sep 23. PMID 26398594
- [Background] Gajewska-Wozniak O, Skup M, Kasicki S, Ziemlinska E, Czarkowska-Bauch J. Enhancing proprioceptive input to motoneurons differentially affects expression of neurotrophin 3 and brain-derived neurotrophic factor in rat hoffmann-reflex circuitry. PLoS One. 2013 Jun 11;8(6):e65937. doi: 10.1371/journal.pone.0065937. Print 2013. PMID 23776573
- [Background] Yamaguchi T, Tanabe S, Watanabe T, Muraoka Y. Effect of voluntary contraction with electrical stimulation to antagonist muscle on agonist H-reflex. Electromyogr Clin Neurophysiol. 2007 Jul;47(4-5):251-5. PMID 17711043
- [Derived] Matsuse H, Segal NA, Rabe KG, Shiba N. Effect of Neuromuscular Electrical Stimulation During Walking on Pain Sensitivity in Women With Obesity With Knee Pain: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 Sep;103(9):1707-1714. doi: 10.1016/j.apmr.2022.01.157. Epub 2022 Mar 23. PMID 35337843
- [Derived] Matsuse H, Segal NA, Rabe KG, Shiba N. The Effect of Neuromuscular Electrical Stimulation During Walking on Muscle Strength and Knee Pain in Obese Women With Knee Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2020 Jan;99(1):56-64. doi: 10.1097/PHM.0000000000001319. PMID 31592880

RESULTS

PARTICIPANT FLOW:
Groups:
- Hybrid Training System (HTS): HTS stimulation while walking at a comfortable pace for 30 minutes.
  Hybrid Training System (HTS): Electrodes will be placed over the quadriceps and hamstrings. Electrical stimulation parameters will be based on a standard Russian waveform in which a 5000 Hz carrier frequency is modulated at 40 Hz (2.4 ms on, 22.6 ms off) to deliver a rectangular voltage biphasic pulse. Acceleration sensors as a joint motion sensor is placed on the front of each leg 88mm above the patellar edge. It analyzes the algorithm of each exercise pattern, and stimulates the antagonist of the motion of each bilateral knee joint during exercise. Electrical stimulation intensity will be set to ~50-60% of 1RM based on the subject's tolerance. The subject's tolerance gradually increases, and electrical stimulation intensity is reset every 2 weeks.
Period: Overall Study
Arm/Group | Hybrid Training System (HTS) | Transcutaneous Electrical Nerve Stimulation (TENS)
Started | 14 | 14
Completed | 10 | 10
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Unrelated Injury affecting outcomes. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hybrid Training System (HTS) | Transcutaneous Electrical Nerve Stimulation (TENS) | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.21 (10.02) | 58.29 (6.35) | 58.75 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kilograms (kg)] — Digital physicians scale (Detecto 6449 Digital Physician Scale, DETECTO Scale Company, Webb City, MO).
  kilograms (kg) | 97.1 (9.6) | 95.6 (12.6) | 96.4 (11.1)
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Wall mounted stadiometer (seca 216 Stadiometer, seca Corporation, Chino, CA)
  centimeters (cm) | 161.5 (6.6) | 163.5 (8.6) | 162.5 (7.6)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meters squared (kg/m2)] — BMI was calculated by dividing body mass by the square of the height.
  kilograms per meters squared (kg/m2) | 37.4 (4.2) | 35.8 (2.9) | 36.6 (3.6)
20-Meter Walk Time [Mean (Standard Deviation); unit: seconds] | 12.5 (2.0) | 12.9 (2.0) | 12.7 (2.0)
5-Chair Stand Time [Mean (Standard Deviation); unit: seconds] | 11.9 (3.1) | 15.2 (4.6) | 13.6 (3.8)
Stair Climb Time [Mean (Standard Deviation); unit: seconds] | 6.4 (1.3) | 6.7 (2.5) | 6.5 (1.9)
Knee Extension Torque [Mean (Standard Deviation); unit: Newton-meters (Nm)] — Maximum isokinetic torque measured on the HUMAC NORM (Model 502140, Computer Sports Medicine, Inc., Stoughton, MA).
  Newton-meters (Nm) | 79.6 (35.9) | 71.7 (42.2) | 75.6 (39.1)
Knee Flexion Torque [Mean (Standard Deviation); unit: Newton-meters (Nm)] — Maximum isokinetic torque measured on the HUMAC NORM (Model 502140, Computer Sports Medicine, Inc., Stoughton, MA).
  Newton-meters (Nm) | 36.8 (22.0) | 26.3 (19.2) | 31.6 (20.6)
Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain Subscale [Mean (Standard Deviation); unit: units on a scale] — The Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain subscale was used at baseline and follow-up to assess participant outcomes. The pain subscale is made up of 9 questions and was scored from zero to 100, with zero corresponding to extreme knee problems and 100 corresponding to no knee problems.
  units on a scale | 14.7 (4.7) | 17.1 (4.0) | 15.9 (4.4)
Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QOL) sub scale [Mean (Standard Deviation); unit: units on a scale] — The Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QOL) subscale was used at baseline and follow-up to assess participant outcomes. The QOL subscale is made up of 4 questions and was scored from zero to 100, with zero corresponding to extreme knee problems and 100 corresponding to no knee problems.
  units on a scale | 9.1 (2.6) | 10.4 (3.0) | 9.8 (2.8)
Knee Pain by Visual Analog Scale [Mean (Standard Deviation); unit: millimeters (mm)] — Knee pain will be evaluated using a visual analog scale (VAS) of 100 mm from no pain (0 mm) to the worst imaginable pain (100 mm). Participants will be asked to record their pain levels of the one week prior to their baseline visit.
  millimeters (mm) | 31.6 (23.4) | 43.6 (22.2) | 37.6 (22.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Extensor Strength Assessed by Isokinetic Dynamometer.
Description: Participants will be familiarized with strength testing equipment and counseled on proper lifting technique. They will undergo testing to determine their peak isokinetic knee extensor torque, using an isokinetic dynamometer.
Time Frame: Baseline and 12-week follow-up
Measure: Least Squares Mean (Standard Error); unit: Newton-meters (Nm)
Arm/Group | Hybrid Training System (HTS) | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 10 | 10
Newton-meters (Nm) | 9.6 (10.8) | 3.8 (28.9)

2. Secondary Outcome: Change in Knee Flexor Strength Assessed by Isokinetic Dynamometer
Description: Participants will be familiarized with strength testing equipment and counseled on proper lifting technique. They will undergo testing to determine their peak isokinetic knee flexor torque, using an isokinetic dynamometer.
Time Frame: Baseline and 12-week follow-up
Measure: Mean (Standard Deviation); unit: Newton-meters (Nm)
Arm/Group | Hybrid Training System (HTS) | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 10 | 10
Newton-meters (Nm) | 9.3 (9.7) | 6.3 (15.1)

3. Secondary Outcome: Change in Knee Pain Assessed by a Visual Analog Scale (VAS)
Description: Knee pain will be evaluated using a visual analog scale (VAS) of 100 mm from no pain (0 mm) to the worst imaginable pain (100 mm). Participants will be asked to record their pain levels of the past one week.
Time Frame: Baseline and 12-week follow-up
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Arm/Group | Hybrid Training System (HTS) | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 10 | 10
millimeters (mm) | -14.9 (27.1) | -11.9 (23.1)

4. Secondary Outcome: Change in Knee Pain Assessed by Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain subscale was used at baseline and follow-up to assess participant outcomes. The pain subscale is made up of 9 questions and was scored from zero to 100, with zero corresponding to extreme knee problems and 100 corresponding to no knee problems.
Time Frame: Baseline and 12-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hybrid Training System (HTS) | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 10 | 10
units on a scale | -5.4 (4.0) | -5.3 (4.9)

5. Secondary Outcome: Change in Quality of Life (QOL) Assessed by Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life (QOL) subscale was used at baseline and follow-up to assess participant outcomes. The QOL subscale is made up of 4 questions and was scored from zero to 100, with zero corresponding to extreme knee problems and 100 corresponding to no knee problems.
Time Frame: Baseline and 12-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hybrid Training System (HTS) | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 10 | 10
units on a scale | -2.6 (1.9) | -2.4 (3.0)

6. Secondary Outcome: Change in 20-meter Walk Time.
Description: Average time of two trials used for each participant.
Time Frame: Baseline and 12-week follow-up
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Hybrid Training System (HTS) | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 10 | 10
seconds | -0.53 (0.9) | -0.52 (1.5)

7. Secondary Outcome: Change in 5-chair Stand Time.
Description: Average time of two trials used for each participant.
Time Frame: Baseline and 12-week follow-up
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Hybrid Training System (HTS) | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 10 | 10
seconds | -1.5 (1.5) | -2.4 (2.9)

8. Secondary Outcome: Change in Stair Climb Time.
Description: Average time of two trials used for each participant.
Time Frame: Baseline and 12-week follow-up
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Hybrid Training System (HTS) | Transcutaneous Electrical Nerve Stimulation (TENS)
Number analyzed (Participants) | 10 | 10
seconds | -0.8 (0.5) | -1.4 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of the study from baseline to 12-week follow-up.
Arm/Group | Hybrid Training System (HTS) | Transcutaneous Electrical Nerve Stimulation (TENS)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 2/14 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hybrid Training System (HTS) (N=14) | Transcutaneous Electrical Nerve Stimulation (TENS) (N=14)
Increased Knee Pain during Intervention (Musculoskeletal and connective tissue disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
The number of participants was insufficient to detect a statistically significant improvement in knee pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-02-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT02730598/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-12-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT02730598/Prot_SAP_001.pdf